CLINICAL TRIAL: NCT00881933
Title: Phase I/II Study of Fludarabine, Cyclophosphamide Plus TBI Conditioning Regimen for Double Units Cord Blood Transplantation in Severe Aplastic Anemia
Brief Title: Study of Fludarabine + Cyclophosphamide + TBI Conditioning Regimen for Double Units Cord Blood Transplantation(CBT)in Severe Aplastic Anemia(SAA)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Korean Society of Pediatric Hematology Oncology (Network)
Responsible Party: The Korean Society of Hematology, The Korean Society of Pediatric Hematology Oncology
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSPHO-SCT0804
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Aplastic Anemia
Keywords: Fludarabine, Cyclophosphamide, TBI, severe aplastic anemia,; cord blood transplantation, pediatric
MeSH Terms: conditions — Anemia, Aplastic; Brain Injuries, Traumatic | interventions — Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine (Experimental)
  Interventions: Other: Cyclophosphosphamide, TBI

INTERVENTIONS:
Other: Cyclophosphosphamide, TBI — fludarabine (30 mg/m2 once daily i.v. on days -7, -6, -5, -4, -3, & -2) (if body weight < 10 kg or if age < 1 year: 1.33 mg/kg) cyclophosphamide (60 mg/kg once daily i.v. on days -9, & -8) total body irradiation (3G on days -1)

SUMMARY:
Severe aplastic anemia is a fatal disease and patients without HLA matched siblings need alternative treatment option. Cord blood transplantation (CBT) has become an alternative treatment means in various diseases, but it has not been proved to be good for severe aplastic anemia. Double units CBT is proposed to have better engraftment potential and and we reported successful double units UCBT after engraftment failure with single unit with promising result. To increase the engraftment potential, fludarabine, cyclophosphamide plus TBI conditioning regimen for double units cord blood transplantation was proposed for the patient with severe aplastic anemia without HLA-matched donor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe aplastic anemia defined by any two or three peripheral blood criteria and either marrow criterion.
* Peripheral blood

  * Neutrophils < 0.5 x 109/l
  * Platelets < 20 x 109/l
  * Corrected reticulocytes < 1%
* Bone marrow

  * Severe hypocellularity (< 25%)
  * Moderate hypocellularity (25-30%) with hematopoietic cells representing < 30% of residual cells
* No prior hematopoietic stem cell transplantation.
* Age: no limits.
* Performance status: ECOG 0-2.
* Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

  * Heart: a shortening fraction > 30%, ejection fraction > 45%.
  * Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
  * Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
* Patients must lack any active viral infections or active fungal infection.
* No appropriate donor
* Appropriate cord blood is available: matched at least in 4/6 of A, B, DR loci.
* Patients (or one of parents if patients age < 19) should sign informed consent.

Exclusion Criteria:

* Pregnant or nursing women.
* Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
* Psychiatric disorder that would preclude compliance.
* Congenital aplastic anemia including Fanconi anemia.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the engraftment potential of fludarabine, busulfan plus thymoglobulin conditioning regimen for cord blood transplantation (CBT) in severe aplastic anemia. | From Oct 2008. to Sep 2011

SECONDARY OUTCOMES:
To evaluate the incidence and severity of toxicity and treatment related mortality | From Oct 2008. to Sep 2011
To evaluate overall and event free survival rate | From Oct 2008. to Sep 2011
To evaluate acute and chronic GVHD | From Oct 2008. to Sep 2011
To evaluate immunologic recovery after CBT | From Oct 2008. to Sep 2011

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Seop Ahn, M.D, Ph.D, Principal Investigator — The Korean Society of Pediatric Hematology Oncology
Locations (1):
- Seoul National University Hospital, Seoul, South Korea